CLINICAL TRIAL: NCT02804659
Title: Physiopathological and Therapeutic Value of microRNA in the Progression of Carotid Artery Plaques: Carotid Protocol and microRNA
Acronym: CAMIA2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2014_843_0024
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Carotid Arteries
Keywords: micro-RNA
MeSH Terms: interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — carotid artery plaques blood

INTERVENTIONS:
Other: microRNA — Extraction of the microRNA using the mirVana miRNA isolation kit and quantification using real-time PCRs

SUMMARY:
Molecular analysis of the atheroma plaque. Screening for a novel biomarker of carotid status.

ELIGIBILITY:
Inclusion Criteria:

* Adults having to undergo carotid thromboendarteriectomy
* social security coverage
* provision of study information
* consent to participation.

Exclusion Criteria:

* Previous carotid artery surgery
* refusal to participate in the study
* or inability to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults having to undergo carotid thrombendarteriectomy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-07; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
expression level of the seven miRNAs of interest | Day of surgery
  expression level of the seven miRNAs of interest in the serum and in carotid artery plaques : miR-100, miR-125a, miR-127, miR-133a, miR-145, miR-221

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MAITRIAS, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France